CLINICAL TRIAL: NCT04996381
Title: Feasibility of Artificial Intelligence-based Heart Function Prediction Model Using Chest Radiography
Brief Title: Feasibility of AI-based Heart Function Prediction Model Using CXR
Acronym: AI-CXR
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Principal Investigator, SungA Bae, MD. PhD., Yonsei University
Other Study IDs: YonseiU
Record Dates: First submitted 2021-08-04; First posted 2021-08-09 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: Chest X-ray for Clinical Evaluation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Scanning Chest X-rays and performing AI algorithms on images — Chest X-Rays; AI CNNs; Results

SUMMARY:
The investigators will develop an artificial intelligence model to predict left ventricular ejection fraction using chest radiographic images and transthoracic echocardiography data.

DETAILED DESCRIPTION:
Echocardiography should be considered at an early stage in patients who have first developed heart failure or who do not have information about heart function, but the examination may be delayed due to lack of time and manpower in the actual medical field.

Primary Objective: Use chest radiographs to predict the left ventricular ejection fraction

ELIGIBILITY:
Inclusion Criteria:

* Adults who are 20 years and older
* Patient who visited the emergency room or outpatient clinic due to dyspnea and chest pain

Exclusion Criteria:

* Patient refusal
* Uncertain radiographs or transthoracic echocardiography
* Uncertain tests results

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing a transthoracic echocardiogram will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 505 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Left Ventricular Ejection Fraction < 40% | Within two weeks of chest X-ray
  Evaluate the performance of chest X-ray based artificial intelligence algorithms to identify individuals with reduced ejection fraction (<40%)

CONTACTS AND LOCATIONS:
Overall Officials: In Hyun Jung, MD, PhD, Study Chair — Yongin Severance Hospital, Yonsei University College of Medicine
Locations (1):
- Yongin Severance Hospital, Yŏngin, Giheung-gu, South Korea